CLINICAL TRIAL: NCT05477589
Title: A Randomized, Multi-Center Phase III Trial Comparing Two Conditioning Regimens (CloFluBu and BuCyMel) in Children With Acute Myeloid Leukemia Undergoing Allogeneic Stem Cell Transplantation.
Brief Title: Studying Conditioning Regimen In Pediatric Transplantation - AML , SCRIPT-AML
Acronym: SCRIPT-AML
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2021-003282-36
Record Dates: First submitted 2022-07-13; First posted 2022-07-28 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-11

CONDITIONS: Acute Myeloid Leukemia (AML) in Remission; Stem Cell Transplantation
Keywords: Leukemia; Leukemia, Myeloid, Acute; Neoplasms; Haematopoietic cell transplantation; Paediatric
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia; Neoplasms | interventions — Busulfan; Cyclophosphamide; Melphalan; Clofarabine; fludarabine

STUDY DESIGN:
Intervention Model Description: AML patient eligible for stem cells transplantation will be randomized either get conditioning regimens CloFluBu or BuCyMel.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BuCyMel (Active Comparator): a combination of busulfan, cyclophosphamide and melphalan, conditioning regimen
  Interventions: Drug: busulfan, cyclophosphamide and melphalan, BuCyMel
- CloFluBu (Experimental): a combination of clofarabine, fludarabine and busulfan conditioning regimen
  Interventions: Drug: clofarabine, fludarabine and busulfan, CloFluBu

INTERVENTIONS:
Drug: busulfan, cyclophosphamide and melphalan, BuCyMel — a three alkylator combination of busulfan, cyclophosphamide and melphalan (BuCyMel, standard arm)
  Other Names: BuCyMel
  Arms: BuCyMel
Drug: clofarabine, fludarabine and busulfan, CloFluBu — combination of clofarabine, fludarabine and busulfan in which two alkylators are replaced by antimetabolites (CloFluBu, experimental arm)
  Other Names: CloFluBu
  Arms: CloFluBu

SUMMARY:
It is a randomized phase 3 study comparing two conditioning regimens in children with Acute Myeloid Leukemia, AML, undergoing allogenic stem cell transplantation. The primary aim is to investigate if a conditioning regimen containing one alkylator (Bu) combined with two antimetabolites (Clo and Flu) results in superior 2-year acute grade III to IV-free, chronic non-limited GvHD-free, relapse free survival than a conditioning regimen combining three alkylating agents (BuCyMel)

DETAILED DESCRIPTION:
The study is designed as an open-label randomized phase III, multicenter superiority trial comparing two conditioning regimens CloFluBu and BuCyMel in children with acute myeloid leukemia (AML) with per-protocol indications to allogeneic hematopoietic stem cell transplantation with a myeloablative conditioning.

This study is composed of two parts - an interventional part that includes randomization, and an observational part. The interventional part is a phase III randomized, open label, multicenter parallel group trial comparing two conditioning regimens used in pediatric HCT: a three alkylator combination of busulfan, cyclophosphamide and melphalan (BuCyMel, standard arm) and a combination of clofarabine, fludarabine and busulfan in which two alkylators are replaced by antimetabolites (CloFluBu, experimental arm). The observational part will prospectively register outcome measures of transplantation in patients not fulfilling criteria for participation in the interventional part of the study (due to lack of complete remission, lack of matched sibling or unrelated donor, who were not recruited to a national upfront protocol or who decline participation in randomization) but consenting to registration of the data.

ELIGIBILITY:
Inclusion criteria for randomization part of the study:

* Age ≤18 years at time of initial AML, age ≤ 21 years at transplantation.
* HCT is performed in a study participating center
* All women of childbearing potential who have to have a negative pregnancy test within 2 weeks prior to the start of treatment.
* Signed informed consent.
* Any relapsed AML after initial treatment according to a defined international AML protocol. (NOPHO-DBH AML 2012/new protocol), or AML in first remission with transplant indications and treatment according to national AML protocol (NOPHO-DBH AML 2012 or new protocol).
* In hematological remission, defined as:

< 5 % leukemic blasts confirmed by flow cytometry (in patients with an informative leukemia associated immunophenotype) in a bone marrow sample taken ≤14 days prior to start of conditioning and no evidence of extramedullary disease, including in CNS and no leukemic blasts in the peripheral blood (verified by flow cytometry in case immature cells are detected in the peripheral blood differential).

-Patients must have a related or unrelated donor fulfilling any of the following criteria: HLA 10/10 allelic matched, identical, sibling BM donor or HLA 10/10 or 9/10 allelic matched related/unrelated BM or PBSC donor orHLA 5-6/6 unrelated or 6-7-8/8 unrelated Cord Blood (UCB)

Inclusion criteria for observation/registration only:

* Diagnosis of acute myeloid leukemia
* Indication for allogeneic stem cell transplantation, as defined by primary treatment protocol or treating physician.
* Age ≤18 years at time of initial AML, age ≤ 21 years at transplantation.
* Not eligible for randomization, either due to lack of consent or not fulfilling inclusion criteria for interventional part of the study.
* Signed informed consent to prospectively register follow-up data.

Exclusion criteria for the randomization part of the study :

* Diagnosis of myelodysplastic syndrome (MDS).
* Diagnosis of juvenile myelomonocytic leukemia (JMML).
* History of previous malignancy (AML diagnosed as secondary cancer).
* Known diagnosis of Fanconi anemia.
* Prior autologous or allogeneic hematopoietic stem cell transplant.
* Planned prophylactic DLI or other immunotherapeutic interventions after HCT that are not included in the upfront protocol, Planned anti-leukemic medication after HCT that are not included in the upfront protocol
* Known intolerance to any of the chemotherapeutic drugs in the protocol.
* Major organ failure precluding administration of planned chemotherapy.
* Patients with uncontrolled bacterial, viral, or fungal infections (currently taking medication and with progression or no clinical improvement) at time of enrollment.
* Severe concomitant disease that does not allow treatment according to the protocol at the investigator's discretion, e.g. malformation syndromes, cardiac malformations, metabolic disorders, renal impairment (<30% of normal glomerular filtration rate), severe pulmonary, hepatic or cardiac impairment due to toxicity or infection.
* Karnofsky / Lansky score < 50%
* Females who are pregnant (positive serum or urine βHCG) or breastfeeding.
* Females of childbearing potential or men who have sexual contact with females of childbearing potential unwilling to use effective forms of birth control or abstinence for one year after transplantation.
* Subjects unwilling or unable to comply with the study procedures.

Exclusion criteria for the observational part of the study:

* Diagnosis of Myelodysplastic syndrome (MDS).
* Diagnosis of Juvenile myelomonocytic leukemia (JMML).
* Age above 21 years at time of transplantation
* No consent is given to prospectively register outcome data
* Prior autologous or allogeneic hematopoietic stem cell transplant.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 170 (Estimated)
Dates: Start 2022-06-07 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
2-year, acute grade III to IV-free, chronic non-limited GvH-free, relapse-free survival (GREF) | 2 years
  To investigate if a conditioning regimen containing one alkylator (Bu) combined with two antimetabolites (Clo and Flu) results in superior 2-year acute grade III to IV-free, chronic non-limited GvHD-free, relapse free survival (GRFS) than a conditioning regimen combining three alkylating agents (BuCyMel)

SECONDARY OUTCOMES:
Neutrophil and platelet engraftment | 28 days post transplantation
  time to engraftment after stem cells transplantation, in all patients
Primary graft failure | +28 days post transplantation
  The incidence of graft failure defined as neutrophil recovery by day +28 post transplantation
Secondary graft failure | 2 years
  The incidence of secondary graft failure
Cumulative incidence of relapse | 2 years
  The incidence of cumulative incidence of relapse during the first two years after transplantation
The association between pre-HCT MRD and relapse | 2 years
  % of remaining leukemic cells in the last bone marrow sample taken before start of conditioning
Cumulative incidence of transplant-related mortality | 2 years
  The incidence of transplant-related mortality at 2 years
Disease-free survival | 2 years
  Disease-free survival at 2 years
Overall survival | 2 years
  Overall survival at 2 years
Immunological recovery | 2 years
  Immunological recovery of CD3+ and CD4+ cells in peripheral blood
Incidence of grade II-IV and III-IV acute GVHD | +180 days post transplantation
  The incidence of acute GvHD
Incidence of chronic GVHD | 2 years
  The incidence of cGVHD
Incidence of grade ≥ 3 toxicity Sinusoidal Obstruction Syndrome/Veno-Occlusive Disease | + 100 days post transplantation
  The rates of grade ≥ 3 Sinusoidal Obstruction Syndrome/Veno-Occlusive Disease
Incidence of grade ≥ 3 toxicity Engraftment Syndrome (ES) | 2 years
  The incidence of engraftment syndome
Incidence of grade ≥ 3 toxicity Transplant-associated thrombotic microangiopathy (TA-TMA) | 2 years
  The incidence of TA-TMA
Incidence of grade ≥ 3 toxicity Hemorrhagic Cystitis (HC) | 2 years
  The incidence of HC
Incidence of grade ≥ 3 infections | 2 years
  The incidence of grade ≥ 3 infections of bacterial, viral and fungal origin
Health-Related Quality of Life, HRQoL. | 2 years
  HRQoL will be measured at baseline and at certain intervals using the quality of life instrument EQ-5D-Y, (Youth)™which include 2 measurements, the descriptive scale ( i.g. the score 1 is no problems and 3 is a lot of problems) and the VAS scale( 1 is the worst health and 100 is the best health that day).
Transplant-associated hormonal and gonadal late effects | 2 years
  the date of spontaneous puberty, date of spontaneous menarche for female patients and mean testicular volume for male patients, use of hormonal replacement therapy and use of fertility preservation
Nutritional status | 2 years
  BMI in kg/m^2 at baseline and post transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Karin Mellgren, Prof. MD, Study Chair — Sahlgrenska University Hospital; Birgitta Versluys, MD, Phd, Principal Investigator — Princess Máxima Center for Pediatric Oncology, Utrecht, The Netherlands
Locations (17):
- Belgium (5):
  - L'Hôpital Universitaire des Enfants Reine Fabiola (HUDERF), Brussels
  - Cliniques Universitaires Saint-Luc (CUSL), Brussels
  - Department of Pediatric Hematology, Oncology and SCT, Ghent University Hospital, Ghent
  - University Hospital Leuven, Leuven
  - Centre Hospitalier Régional de la Citadelle (CHR)/CHU Liège, Liège
- Paediatric Stem Cell Transplant and Immune Deficiency, Department of Pediatric and Adolescent Medicine, Section 4072, Rigshospitalet University Hospital of Copenhagen, Copenhagen, Denmark
- Division of Hematology, Oncology, and Stem Cell Transplantation, The New Children's Hospital, Helsinki University Hospital, Helsinki, Finland
- Department of Pediatrics and Adolescent Medicine, Hong King Children's Hospital, Hong Kong, Hong Kong
- Schneider Children's Medical Center of Israel, Petah Tikva, Israel
- Vilnius University Hospital Santaros Klinikos Center for Pediatric Oncology and Hematology, Vilnius, Lithuania
- Princess Máxima Center for Pediatric Oncology, Utrecht, Netherlands
- Department of Pediatric Hematology and Oncology, Oslo University HospitalOslo University Hospital, Oslo, Norway
- Stemcelltransplant unit Hospital Niño Jesús, Madrid, Spain
- Sweden (4):
  - Queen Silvia Children's Hospital, Sahlgrenska University Hospital, Gothenburg
  - Barncancercentrum, avdelning 64, Skane University Hospital, Lund
  - Pediatric Hematology immunology and stem cell transplantation Astrid Lindgren children's Hospital Huddinge K86-88, Stockholm
  - Childrens department for Blood and tumor diseases Uppsala University Hospital, Uppsala